CLINICAL TRIAL: NCT02924259
Title: Does Self-myofascial Release With a Foam Roll Change Pressure Pain Threshold of the Ipsilateral Lower Extremity Agonist, Antagonist, and Contralateral Muscle Groups? an Exploratory Study
Brief Title: Does Self-myofascial Release With a Foam Roll Change Pressure Pain Thresholds in Lower Extremity Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Dominguez Hills (Other)
Responsible Party: Principal Investigator, Scott Cheatham, Assistant Professor, California State University, Dominguez Hills
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.17-039
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Myofascial Pain Syndromes
Keywords: muscle soreness; pain; myofascial release
MeSH Terms: conditions — Myofascial Pain Syndromes; Myalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foam Roll Group (Experimental): Subjects will undergo a 2-minute video-guided foam roll intervention on the left quadriceps muscle using the GRID foam roll.
  Interventions: Device: The GRID foam roll

INTERVENTIONS:
Device: The GRID foam roll — Commercial rigid foam roll with an outer foam covering

SUMMARY:
The purpose of this study was to examine the effects of a foam rolling intervention on pressure pain thresholds (PPT) of the ipsilateral antagonist and contralateral muscle groups. Through this research we sought to gather data to further develop the methodology for future studies of this intervention.

DETAILED DESCRIPTION:
To date, no studies have examined how foam rolling effects the PPT of the ipsilateral antagonist and contralateral muscle. There is a gap in the literature regarding our knowledge of the effects of foam rolling on these muscles. This will be the first study to examine the acute effects of a foam rolling intervention on ipsilateral antagonist and contralateral muscle group PPT.

Forty-five (N=45) healthy adults (18-65 years) from California State University Dominguez Hills (CSUDH) will be recruited for this study via convenience sampling. Data collection will take place in the CSUDH sports medicine laboratory. Prior to testing, participants will fill out a screening questionnaire with questions that represent the exclusion criteria which will be used to determine ineligibility for this study.

Prior to participant recruitment and enrollment, a pilot study will be done on 10 participants to establish rater reliability using the methods mentioned below. After acceptable reliability is achieved, recruitment and enrollment will continue.

Participants who meet the inclusion criteria and consent to participate will be enrolled in the study. Participants will read and sign a CSUDH approved consent form prior to beginning data collection. Following consent, participants will also fill out a questionnaire to provide demographic information which includes age, height, and weight.

Following completion of the paperwork, all participants will undergo testing which will be conducted between the hours of 10am and 2pm. Each data collection session will last for approximately 10 minutes. Pressure pain threshold (PPT) will be measured using a digital algometer on the ipsilateral left quadriceps, left hamstring, and right quadriceps muscle group. All subjects will follow a 2-minute video-guided foam roll intervention on the left quadriceps using a rigid foam roll with outer foam covering. The data collection process is as follows:

1. Pretest measures (subject standing): PPT of the ipsilateral left quadriceps, left hamstring and right quadriceps group (subject is standing during testing)
2. Intervention: 2-minute video-guided foam roll intervention using a rigid foam roller.
3. Posttest measures (subject standing): PPT of the ipsilateral left quadriceps, left hamstring, and right quadriceps group.

Collected data will be transferred to SPSS v.22 (IBM SPSS, Chicago, IL). Means,standard deviations, 95% confidence intervals (95% CI), and ranges for participant descriptive data will be calculated. Pressure pain threshold pretest and posttest differences will be calculated using the paired t-test The p-value will be considered significant at the .05 level using a two-tailed test (α2 =.05)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Musculoskeletal, systemic, or metabolic disease that would affect lower extremity joint ROM or tolerance to pressure pain threshold testing and the inability to avoid medications that may affect testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline pressure pain threshold to immediate post intervention. | baseline and immediately post intervention
  Pressure pain threshold will be tested immediately before the intervention and immediately after the intervention on the left hamstring and right quadriceps muscle groups.

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Cheatham, PhD, DPT, Principal Investigator — CSUDH
Locations (1):
- Cal State University Dominguez Hills, Carson, California, United States

IPD SHARING:
Plan to Share IPD: No